CLINICAL TRIAL: NCT07213245
Title: Metabolic Effects of Short-term Ultra-processed Food Intake (MEST-UPF): a Randomized Controlled Trial
Brief Title: Metabolic Effects of Short-term Ultra-processed Food Intake (MEST-UPF)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: MEST-UPF
Record Dates: First submitted 2025-09-23; First posted 2025-10-08 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-11

CONDITIONS: Appetite; Obesity and Obesity-related Medical Conditions
MeSH Terms: conditions — Obesity | interventions — Food, Processed

STUDY DESIGN:
Intervention Model Description: Factorial assignment 2X2 factorial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Meal high in energy density, high in ultra-processed food (Experimental): Meal high in energy density, high in ultra-processed food
  Interventions: Other: Meal high in energy density, high in ultra-processed food
- Meal high in energy density, low in ultra-processed food (Experimental): Meal high in energy density, low in ultra-processed food
  Interventions: Other: Meal high in energy density, low in ultra-processed food
- Meal low in energy density, high in ultra-processed food (Experimental): Meal low in energy density, high in ultra-processed food
  Interventions: Other: Meal low in energy density, high in ultra-processed food
- Meal low in energy density, low in ultra-processed food (Experimental): Meal low in energy density, low in ultra-processed food
  Interventions: Other: Meal low in energy density, low in ultra-processed food

INTERVENTIONS:
Other: Meal high in energy density, high in ultra-processed food — Meal high in energy density, high in ultra-processed food
  Arms: Meal high in energy density, high in ultra-processed food
Other: Meal high in energy density, low in ultra-processed food — Meal high in energy density, low in ultra-processed food
  Arms: Meal high in energy density, low in ultra-processed food
Other: Meal low in energy density, high in ultra-processed food — Meal low in energy density, high in ultra-processed food
  Arms: Meal low in energy density, high in ultra-processed food
Other: Meal low in energy density, low in ultra-processed food — Meal low in energy density, low in ultra-processed food
  Arms: Meal low in energy density, low in ultra-processed food

SUMMARY:
The overall aim of this project is to study the effects of short-term high ultra-processed food intake, compared to nutrient- and energy density matched low ultra-processed food (UPF) intake, on energy intake and appetite.

A total of 24 men and women who meet all inclusion criteria and none of the exclusion criteria will be invited to participate. A randomized 2*2 factorial four-way crossover study will be conducted at the Department of Internal medicine and Clinical Nutrition at the University of Gothenburg, comparing a high-UPF meal to a low-UPF meal also with high and/or low energy density. A supervised breakfast meal will be served, and postprandial blood samples and appetite measures will be collected continuously up to 4 hours after the breakfast meal. Subsequently, an ad libitum lunch meal will be served, and energy intake will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) 18.5-30 kg/m2
* Fasting glucose < 6.1 mmol/l
* Hb >110 g/L
* Weight stability the last 3 months +/-5%

Exclusion Criteria:

* Food allergies, intolerances or preferences preventing consumption of any products included in the study.
* Unable to sufficiently understand written and spoken Swedish or English to provide written consent and understand information and instructions from the study personal.
* Pregnant, lactating or planning a pregnancy during the study period.
* Blood donation or participation in a clinical study with blood sampling within 30 days prior to screening visit and throughout the study.
* History of gastrointestinal conditions or major gastrointestinal surgery (Inflammatory bowel disease, Crohn's disease, malabsorption, colostomy, bowel resection, gastric bypass surgery etc.).
* Type 1 diabetes or type 2 diabetes.
* Thyroid disorder.
* Current smoking, vaping.
* Following any weight reduction program or having followed one during the last 6 months prior to screening.
* Not habitually eating breakfast (<5 times/week).
* Restrained eating based on the three-factor eating questionnaire.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Self-reported appetite | Baseline to 8 hours after test meal
  Appetite ratings (hunger, fullness, and desire to eat) will be assessed using separate 100-mm Visual Analogue Scales (VAS), anchored with "not at all" (0 mm) and "extremely" (100 mm). Higher scores indicate greater perceived intensity.
Energy intake | 4 hours after test meal
  Energy intake estimated by nutrient calculation of leftover food at the ad libitum lunch meal
Gastrointestinal hormones - incretins | Baseline to 4 hours after test meal
  Difference between groups in incretins GIP and GLP-1 in response to meal
Gastrointestinal hormones - cholecystokinin | Baseline to 4 hours after test meal
  Difference between groups in cholecystokinin in response to meal
Gastrointestinal hormones - peptide YY | Baseline to 4 hours after test meal
  Difference between groups in peptide YY (PYY) in response to meal
Gastrointestinal hormones - ghrelin | Baseline to 4 hours after test meal
  Difference between groups in ghrelin in response to meal

SECONDARY OUTCOMES:
Eating rate | Baseline til end of study meal
  Time it takes to eat the study meal until satisfied
Glucose postprandial | Baseline to 4 hours after test meal
  Difference between groups in postprandial glucose in response to meal.
Insulin postprandial | Baseline to 4 hours after test meal
  Difference between groups in postprandial insulin in response to meal.
Lipid metabolism | Baseline to 4 hours after test meal
  Difference between groups in postprandial lipid metabolism in response to meal.
Metabolome | Baseline to 4 hours after test meal
  Differences between groups in metabolome (plasma) measured using metabolomics in response to meals.
Proteome | Baseline to 4 hours after test meal
  Differences between groups in proteome (plasma) measured using proteomics in response to meals.
Self-reported prospective energy intake | From 30 min until midnight or bedtime (which ever comes first)
  Self-reported prospective energy intake during the remainder of the day
Inflammatory markers in blood - cytokines | Baseline to 4 hours after test meal
  Differences between groups in immunological responses (cytokines) in response to meal.
Inflammatory markers in blood - lipopolysaccharides | Baseline to 4 hours after test meal
  Differences between groups in immunological responses (lipopolysaccharides) in response to meal.
Inflammatory markers in blood - GlycA | Baseline to 4 hours after test meal
  Differences between groups in immunological responses (GlycA) in response to meal.
Lipid profile | Baseline to 4 hours after test meal
  Differences between groups in lipid profile (plasma) measured using lipidomics in response to meals.

OTHER OUTCOMES:
Determinants of energy intake - proteome | Baseline
  Correlation between baseline proteome measured using proteomics and the primary outcome energy intake
Determinants of energy intake - metabolome | Baseline
  Correlation between baseline metabolome measured using metabolomics and primary outcome energy intake
Determinants of energy intake - body composition | Baseline
  Correlation between baseline body composition (fat percentage and fat free mass percentage) measured using Bioelectrical impedance analysis (BIA) and primary outcome energy intake
Determinants of energy intake - metabolic markers | Baseline
  Correlation between baseline metabolic markers, fasting plasma glucose, insulin, and triglycerides measured via standard clinical chemistry methods, and primary outcome energy intake
Determinants of energy intake - physical activity | Baseline
  Correlation between baseline self-reported physical activity and primary outcome energy intake
Determinants of energy intake - diet | Baseline
  Correlation between baseline diet (macro- and micronutrient intake, dietary patterns, food group intake) estimated from a 4-day dietary record and primary outcome energy intake
Determinants of energy intake - microbiome | Baseline
  Correlation between baseline gut microbiome composition-assessed using metagenomic shotgun sequencing and 16S rRNA analysis-and the primary outcome of energy intake.

CONTACTS AND LOCATIONS:
Overall Officials: Therese Karlsson, PhD, Principal Investigator — University of Gothenburg, Institute of medicine
Locations (1):
- Department of internal medicine and clinical nutrition, University olf Gothenburg, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Undecided